CLINICAL TRIAL: NCT03757351
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL747 in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Study to Evaluate DNL747 in Subjects With Amyotrophic Lateral Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to change in Sanofi's development strategy for DNL747/SAR443060 - not due to any safety concerns
Sponsor: Sanofi (Industry)
Collaborators: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TDR16536; DNLI-D-0003 (Other: Denali Therapeutics Inc.)
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- DNL747 First, Placebo Second (Experimental)
  Interventions: Drug: DNL747; Drug: Placebo
- Placebo First, DNL747 Second (Experimental)
  Interventions: Drug: DNL747; Drug: Placebo
- Open-Label Extension (Experimental): Conducted in the Netherlands only.
  Interventions: Drug: DNL747

INTERVENTIONS:
Drug: DNL747 — Repeating oral dose
Drug: Placebo — Repeating oral dose
  Arms: DNL747 First, Placebo Second; Placebo First, DNL747 Second

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple oral doses of DNL747 in subjects with Amyotrophic Lateral Sclerosis in a cross-over design

ELIGIBILITY:
Key Inclusion Criteria (Double-Blind Part):

* Women of non-childbearing potential and men, aged 21-80 years
* Willingness and ability to complete all aspects of the study; participant should be capable of completing assessments either alone or with help of a caregiver
* Diagnosis of laboratory-supported probable, probable, or definite (sporadic or familial) ALS according to the El Escorial World Federation of Neurology revised research diagnostic criteria
* Less than 3 years since symptom onset
* Forced vital capacity (FVC) >50% predicted measured within 30 days of screening
* If subject is taking approved ALS treatments (riluzole and/or edaravone), doses must be stable for ≥2 months prior to screening and subject is expected to stay on a stable regimen throughout the study

Key Exclusion Criteria (Double-Blind Part):

* History of a clinically significant non-ALS neurologic disorder (other than frontal temporal lobe dementia), including, but not limited to, muscular dystrophy, spinal stenosis, peripheral neuropathy, inherited neuropathies, AD, Parkinson's disease, Lewy body dementia, vascular dementia, Huntington's disease, epilepsy, stroke, multiple sclerosis, brain tumor, or brain infection or abscess
* Unstable or poorly controlled comorbid disease process of any organ system currently requiring active treatment or likely to require treatment adjustment during the study

Key Inclusion Criteria (Open-Label Extension):

* Successful completion of both periods of the the double-blind, crossover part of the study
* Continued diagnosis of laboratory-supported probable, probable, or definite (sporadic or familial) ALS according to the El Escorial World Federation of Neurology revised research diagnostic criteria

Key Exclusion Criteria (Open-Label Extension):

* Presence of laboratory abnormalities, physical examination findings, or AEs determined to be clinically significant by the investigator from the double-blind part of the study that have not resolved by the final follow-up visit as part of the double-blind study period
* New diagnosis of clinically significant neurological disorder (other than frontal temporal lobe dementia)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Randomization - Day 86
Number of Subjects with clinically significant neurological examination abnormalities | Randomization - Day 86
Number of Subjects with laboratory test abnormalities | Randomization - Day 86

SECONDARY OUTCOMES:
Pharmacokinetic measure of maximum observed plasma concentration (Cmax) of DNL747 | Randomization - Day 86
Pharmacokinetic measure of time to reach maximum observed plasma concentration (Tmax) of DNL747 | Randomization - Day 86
Pharmacokinetic measure of area under the plasma drug concentration-time curve (AUC) of DNL747 | Randomization - Day 86
Pharmacokinetic terminal disposition rate constant (λz) with the respective t1/2 of DNL747 | Randomization - Day 86
Pharmacokinetic measure of CSF concentrations of DNL747 | Randomization - Day 86
Pharmacodynamic measure of pS166 in PBMCs | Randomization - Day 86

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (2):
  - Bioclinica, Orlando, Florida
  - PRA Health Sciences, Salt Lake City, Utah
- CHDR, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Vissers MFJM, Heuberger JAAC, Groeneveld GJ, Oude Nijhuis J, De Deyn PP, Hadi S, Harris J, Tsai RM, Cruz-Herranz A, Huang F, Tong V, Erickson R, Zhu Y, Scearce-Levie K, Hsiao-Nakamoto J, Tang X, Chang M, Fox BM, Estrada AA, Pomponio RJ, Alonso-Alonso M, Zilberstein M, Atassi N, Troyer MD, Ho C. Safety, pharmacokinetics and target engagement of novel RIPK1 inhibitor SAR443060 (DNL747) for neurodegenerative disorders: Randomized, placebo-controlled, double-blind phase I/Ib studies in healthy subjects and patients. Clin Transl Sci. 2022 Aug;15(8):2010-2023. doi: 10.1111/cts.13317. Epub 2022 Jun 1. PMID 35649245
- See also: TDR16536 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25354&tenant=MT_SNY_9011